CLINICAL TRIAL: NCT06594198
Title: Evaluation of the BRAINDEX Brain Monitor in Cardiac Surgery, Interventional Comparative Study
Acronym: ARGOS Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Braindex (Industry)
Collaborators: Clinique de la Sauvegarde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A00125
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Brain Monitor; Anaesthesia
Keywords: Brain Monitor; ARGOS Platform; SctO2; ANI; bcSEF; EEG bispectral index; Cerebral tissue oxygen saturation; Analgesia Nociception Index
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Intervention Model Description: Single-centre, prospective, interventional clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One center and 40 patients (Experimental): Monitor the values of 3 brain parameters: SctO2, bcSEF and ANI measured by the ARGOS sensor.
  Interventions: Device: Cerebral monitor

INTERVENTIONS:
Device: Cerebral monitor — The study procedure consists of monitoring the values of 3 cerebral parameters: SctO2, bcSEF and ANI measured by the ARGOS sensor. These 3 parameters will be recorded and compared after the intervention with 3 parameters considered as standard: SctO2 measured by the INVOS 7100 cerebral oximeter, the bispectral index (BIS) measured by the BIS monitor and the ANI measured by the MDoloris monitor. These 3 reference parameters are once again usually monitored and recommended for all cardiac surgery.

SUMMARY:
The main objective of this study is to show the concordance of the SctO2 values of the ARGOS platform with the standard SctO2 values (comparative study with platform INVOS, Medtronic).

DETAILED DESCRIPTION:
SctO2 values from ARGOS and INVOS will be resampled every 30 seconds. The two signals will then be resynchronized and compared on a sample-by-sample basis using a Pearson correlation test. Bias and agreement limits will be assessed using Bland & Altmann graphs. This test will be carried out for the entire duration of the recording.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age
* Patient scheduled for cardiac surgery with programmed extracorporeal circulation (ECC)
* Patient with no history of scalp injury or or skin diseases
* Patient with an Euroscore 2 of less than 7%.
* Patient affiliated or entitled to a social assurance

Exclusion Criteria:

* Weight under 40 kg
* Frontal surface too small to allow application of SctO2, BIS electrodes on the same hemifront
* Patient with severe, unbalanced hypertension
* Measurement of systolic blood pressure (SBP) > 180 mm Hg and/or diastolic blood pressure (DBP) > 110 mm Hg
* Patients undergoing emergency surgery
* Patient with chronic renal failure, with glomerular filtration < 30 ml/min/1.73m², or requiring renal transplantation or requiring renal transplantation
* Patient with left ventricular ejection fraction < 40%
* Patient with a history of ischemic stroke
* Patients with preoperative sepsis
* Patient requiring noradrenaline infusion noradrenaline infusion in the 24 hours prior to surgery
* Patient with preoperative uni or bilateral carotid stenosis bilateral carotid stenosis > 50%.
* Protected patient: adult under guardianship, curatorship or legal protection, deprived of liberty by judicial or administrative decision.
* Pregnant, parturient or breast-feeding women.
* Patients hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Comparison of SctO2 values from ARGOS and INVOS | During the surgical procedure
  Compare ARGOS and INVOS SctO2 values at different times of interest during the procedure.
  Compare ARGOS SctO2 values with invasive central venous and arterial saturation (measured by gasometry) during aortic unclamping.
  Compare INVOS SctO2 values with central venous and arterial saturation before, during and after aortic unclamping.

SECONDARY OUTCOMES:
ANI and Database | During the surgical procedure
  For ANI: Compare the ANI values of the ARGOS device with the ANI values of the reference device (ANIv2 monitor, MDoloris Medical Systems).
  For the bcSEF: Compare the bcSEF values of the ARGOS and the BIS values at different characteristic times during the procedure.
  Build up a database for secondary analysis by continuously recording all data.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No